CLINICAL TRIAL: NCT01492322
Title: Use of SPECT (Single-photon Emission Computed Tomography) to Examine the Role of DAT (Dopamine Transporter) Genotype in Motivated Smoking Behavior
Brief Title: SPECT Imaging of DAT Genotype
Acronym: DDAT
Status: Terminated | Type: Observational
Why Stopped: UPenn suspended production of the ligand necessary to produce the tracer TRODAT.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 813475
Record Dates: First submitted 2011-12-02; First posted 2011-12-14 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2011-12

CONDITIONS: Nicotine Withdrawal
Keywords: Smoker; SPECT; Dopamine; Nicotine Sated condition; Nicotine withdrawal condition

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sated and withdrawal group: To determine differences in TRODAT binding to the DAT between a smoker when sated and when in withdrawal
  Interventions: Radiation: TRODAT

INTERVENTIONS:
Radiation: TRODAT — Smoker will receive a TRODAT injection

SUMMARY:
A polymorphism in the dopamine transporter (DAT) may determine how much dopamine is available at the synapse and this may affect the underlying reasons for relapse in smokers. This research will use Single-photon emission computed tomography SPECT and the DAT-specific ligand, TRODAT (Dopamine Transporter Density by [99mTc]), to examine the availability of DAT in smokers grouped by genotype in the sated (just having smoked) and withdrawal (4 hours without smoking) conditions.

DETAILED DESCRIPTION:
There will be 2 SPECT scans for each smoker who participates in this research. One SPECT scan when the smoker is sated with nicotine and one where the smoker is in withdrawal

ELIGIBILITY:
Inclusion Criteria:

1. Physically healthy male or female nicotine dependent patients ages 18-60 without other current drug dependence (excluding marijuana) or psychiatric diagnosis.
2. Smoke at least 10 cigarettes per day for at least 6 months prior to study start date.
3. Females must be non-pregnant, non-lactating and either be of non-childbearing potential (i.e. sterilized via hysterectomy or bilateral tubal ligation or at least 1 year post-menopausal) or of child bearing potential, but practicing a medically acceptable method of birth control from at least 48 hours prior to SPECT imaging until 30 days following the scan. Examples of medically acceptable methods for this protocol include barrier (diaphragm or condom) with spermicide, an intrauterine device (IUD), oral contraceptives, levonorgestrel implant, or complete abstinence.
4. Subjects provide voluntary informed consent.
5. Subjects must read on 8th grade (or above) level.
6. Not using other methods for smoking cessation

Exclusion Criteria:

1. Participation in clinical trial and receipt of investigational drug(s) during previous 60 days
2. History of head trauma or injury causing loss of consciousness, lasting more than three (3) minutes or associated with skull fracture or inter-cranial bleeding or abnormal MRI.
3. HIV positive on medication for symptoms. This will be determined on an individual basis by results from the physical examination and final approval by our study physician.
4. Symptomatic presence of other hematological disease.
5. Clinically significant cardiovascular, hepatic (liver), renal (kidney), neurological, or endocrinological (including Type II diabetes) abnormalities.
6. Asthmatic condition which requires the use of an inhaler more than twice per week
7. History of psychosis, seizures, or organic brain syndrome.
8. Use of medications or natural herbs that may cause sedation or may effect the brain systems that are being studied (medication use will be evaluated by our study physician on a case-by-case basis).
9. Claustrophobia, trypanophobia (needle phobia) or other medical condition preventing subject from lying in the SPECT scanner for approximately one (1) hour.
10. Individuals with an intelligence quotient of 80 or less.
11. Smoke non-filtered cigarettes
12. Treatment for alcohol or drug dependence within the last 3 months
13. A significant alcohol or drug use history (multiple treatments, 5 years of dependence, positive urines, etc.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects will be forty physically-healthy and mentally-stable male and non-pregnant female subjects between the ages of 18 and 60 who meet the DSM-IV criteria for nicotine dependence. Subjects will not be excluded based on gender, religion, race, or socioeconomic status. The subject population of previous smoking studies in our lab was 54% female, 62% Caucasian, and averaged 15 years of education. This is representative of the urban population in the northeast region of the United States who seek help for nicotine dependence. We expect our current population to have similar characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
SPECT Imaging of DAT Genotype - Difference in TRODAT binding to DAT | Up to 3 years for data analyses
  To determine differences in TRODAT binding to the DAT between smokers who are sated and those who are in withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Franklin, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Addiction Treatment Research Center, Philadelphia, Pennsylvania, United States